CLINICAL TRIAL: NCT02864186
Title: A Randomized Study to Test the Hypothesis That a Support Bra Will Improve Healing and Quality of Life After Coronary Artery By-Pass Graft (CABG)
Brief Title: The Benefits of the Use of a Support Bra in Women Undergoing Coronary Artery By-Pass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Antonio M. Cesar, Associated Professor of Cardiology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDC4123/14/103
Record Dates: First submitted 2016-07-18; First posted 2016-08-11 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Quality of Life; Wound Complications; Pain
Keywords: Pain; Quality of life; wound healing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Active Comparator): Women wont use support bra for six months
  Interventions: Device: control
- surgical support bra (Active Comparator): Women will use surgical support bra 24 hours a day for six months
  Interventions: Device: surgical support bra
- common support bra (Active Comparator): Women will use common support bra 24 hours a day for six months
  Interventions: Device: common support bra

INTERVENTIONS:
Device: control — Women wont use support bra 24 hours a days for six months
  Arms: control
Device: surgical support bra — Women will use surgical support bra 24 hours a day for six months
  Arms: surgical support bra
Device: common support bra — Women will use common support bra 24 hours a day for six months
  Arms: common support bra

SUMMARY:
That study have the primary purpose identify if exist difference to the healing and quality of life between women that use of a surgical support bra, common support bra and without support bra after coronary artery bypass graft surgery.

To do this, will be assessed pain, healing of the wound (dehiscence, infection) and quality of life life through specific instruments.

DETAILED DESCRIPTION:
The patients will be randomized and share into three groups: women after coronary artery bypass surgery use surgical support bra, women after coronary artery bypass surgery use common support bra and those who will not use any support bra.

They will be can tracked and invited to participate in the study few days before the surgery or during the post operatory (2 - 6 days after surgery). The assessement and the intervention must be start in the inpatient unit from the 2nd to 6th post operatory until their discharge.

Initially, it will be apply a questionnaire of quality of life (SF36) to assess the quality of life before the surgical procedure. In this moment, will be measured for breast size and also wil be identify the risk factors through a brief historical.

During the stay in the hospital, the patients will be assessed on a daily basis with respect to the following: pain (verbal numerical scale) and wound appearance.

The questionnaire of quality of life(SF36) will be applied again for more three times, about one month, two months and six months after the discharge together with the assessement to the pain and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergoing coronary artery bypass graft surgery
* Women who signed the term consent and informed

Exclusion Criteria:

* Women who have had any breast surgery
* Women who undergoing radiotherapy to the thorax.
* Women with cognitive impairments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Pain - Visual Numeric Scale - Medical Documentation or Nursing in the Medical | at six months after surgery

SECONDARY OUTCOMES:
Quality of Life pre cardiac surgery - SF36 | one day before surgery and then at one, two and six months
Sternal Wound Dehiscence - Medical Documentation or Nursing in the Medical Records | at six months after surgery
Use of antibiotics and painkillers - Medical Prescription | at six months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: LUIZ AM CESAR, MD, PhD, Principal Investigator — INSTITUTO DO CORAÇÃO, HOSPITAL DAS CLÍNICAS DA FACULDADE DE MEDICINA DA UNIVERSIDADE DE SÃO PAULO
Locations (1):
- Heart Institute (InCor), Univ. of Sao Paulo Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva TRA, Ono JN, Miname FCBR, Gowdak LHW, Mioto BM, Santos RBD, Dallan LRP, Machado Cesar LA. Benefits of using a support bra in women undergoing coronary artery bypass graft surgery: A randomized trial. Clinics (Sao Paulo). 2024 May 20;79:100370. doi: 10.1016/j.clinsp.2024.100370. eCollection 2024. PMID 38772100